CLINICAL TRIAL: NCT01221870
Title: A Phase II Study of Tesetaxel as First-line Therapy for Subjects With Metastatic Breast Cancer
Brief Title: Tesetaxel as First-line Therapy for Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOB203
Record Dates: First submitted 2010-10-13; First posted 2010-10-15 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Breast Neoplasm
Keywords: Metastatic breast cancer; First-line therapy; Tesetaxel; Oral taxane
MeSH Terms: conditions — Breast Neoplasms | interventions — tesetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tesetaxel once every 3 weeks (Experimental): Tesetaxel 27 mg/m2 orally once every 21 days for up to 12 months
  Interventions: Drug: Tesetaxel once every 3 weeks
- Tesetaxel once weekly (Experimental): Tesetaxel 15 mg/m2 orally once every 7 days for 3 consecutive weeks in a 28-day cycle for up to 12 months
  Interventions: Drug: Tesetaxel once weekly

INTERVENTIONS:
Drug: Tesetaxel once every 3 weeks — Tesetaxel capsules orally once every 21 days; duration of therapy not to exceed 12 months
  Other Names: DJ-927
  Arms: Tesetaxel once every 3 weeks
Drug: Tesetaxel once weekly — Tesetaxel capsules orally once every 7 days for 3 consecutive weeks in a 28-day cycle; duration of therapy not to exceed 12 months
  Other Names: DJ-927
  Arms: Tesetaxel once weekly

SUMMARY:
The intravenously administered taxane, paclitaxel, is one of the most commonly employed agents for the treatment of both localized and advanced breast cancer.

Tesetaxel is an orally administered taxane that is in development as first- and second-line treatment for patients with advanced cancers. This study is being undertaken to determine the efficacy and safety of tesetaxel administered as first-line therapy to patients with metastatic breast cancer.

ELIGIBILITY:
Primary Inclusion Criteria:

* Female
* At least 18 years of age
* Histologically or cytologically confirmed adenocarcinoma of the breast
* Stage IV disease
* HER2 status negative
* Measurable disease (revised RECIST; Version 1.1)
* Eastern Cooperative Oncology Group performance status 0 or 1
* Life expectancy of at least 3 months
* Chemotherapy naïve or 1 prior chemotherapy regimen in the adjuvant setting (Prior taxane-based adjuvant therapy allowed provided patient had a disease-free interval of at least 12 months after completing this adjuvant therapy)
* Prior hormonal therapy, aromatase inhibitor therapy, and immunotherapy allowed
* Prior radiotherapy in the adjuvant setting allowed provided that less than 25% of the bone marrow had been irradiated
* Adequate bone marrow, hepatic, and renal function, as specified in the protocol
* At least 4 weeks and recovery from effects of prior surgery, hormonal therapy, aromatase inhibitor therapy, immunotherapy, radiotherapy, or other therapy with an approved or investigational agent
* Ability to swallow an oral solid-dosage form of medication

Primary Exclusion Criteria:

* Known metastasis to the central nervous system
* History of other malignancy within the last 5 years other than curatively treated basal and squamous cell carcinoma of the skin or carcinoma of the cervix in situ
* Significant medical disease other than Stage IV breast cancer
* Presence of neuropathy > Grade 1 (NCI CTC, Version 4.0)
* History of hypersensitivity to a taxane
* Need to continue any regularly-taken medication that is a potent inhibitor or inducer of the CYP3A pathway or P-glycoprotein activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-10 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Response rate (revised RECIST) | 12 months from date of first dose of study medication for last patient enrolled
  Proportion of patients with a confirmed complete or partial response

SECONDARY OUTCOMES:
Disease control rate | 12 months from date of first dose of study medication for last patient enrolled
  Proportion of patients with a confirmed complete or partial response of any duration or stable disease ≥ 3 months in duration
Progression-free rate | 6 months from date of first dose of study medication for last patient enrolled
  Proportion of patients without disease progression 6 months following the first dose of study medication
Durable response rate | 12 months from date of first dose of study medication for last patient enrolled
  Proportion of patients with a confirmed complete or partial response ≥ 6 months in duration
Duration of response | 12 months from date of first dose of study medication for last patient enrolled
  Date when response criteria are first met to the date when progression is first documented
Time to progression | 12 months from date of first dose of study medication for last patient enrolled
  Date of first dose of study medication to the date when progression is first documented
Adverse events | Up to 30 days after the last dose of study medication for a specific patient
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Seidman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The Moses H. Cone Regional Cancer Center, Greensboro, North Carolina
  - The West Clinic, Memphis, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas